CLINICAL TRIAL: NCT03248492
Title: A Phase 2, Multicenter, Open-Label Study of DS-8201a, an Anti-HER2-Antibody Drug Conjugate (ADC) for HER2-Positive, Unresectable and/or Metastatic Breast Cancer Subjects Previously Treated With T-DM1 (DESTINY-Breast01)
Brief Title: A Study of DS-8201a in Metastatic Breast Cancer Previously Treated With Trastuzumab Emtansine (T-DM1)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The last participant was transitioned to alternative study.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); Daiichi Sankyo Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-A-U201; 2016-004986-18 (EudraCT Number); JapicCTI-173693(en) (Registry Identifier: JapicCTI); DESTINY-Breast01 (Other: Daiichi Sankyo and AstraZeneca)
Record Dates: First submitted 2017-08-10; First posted 2017-08-14 (Actual); Results first posted 2020-02-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: HER-2 positive breast cancer; Metastatic or Unresectable; Resistant or refractory to T-DM1; DESTINY - Breast 01; Trastuzumab deruxtecan; T-DXd
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — trastuzumab deruxtecan

STUDY DESIGN:
Intervention Model Description: HER2-positive patients will be classified into two groups: T-DM1 resistant/refractory (experimental) and T-DM1 intolerant (exploratory only).
Masking Description: In Part 1, about 60 trastuzumab emtansine (T-DM1) resistant/refractory patients initially will be randomized into three treatment groups (low, medium and high doses) for Pharmacokinetics (PK), then about another 60 will be randomized into low and high doses to determine recommended dose (RD). After that, about 100 will receive the recommended dose in an open-label continuation stage (Part 2). About 10 TDM-1 intolerant patients will join the continuation stage as an exploratory only arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DS-8201a Low Dose (Experimental): T-DM1 resistant/refractory (R/R) patients in the low dose treatment group
  Interventions: Drug: DS-8201a
- DS-8201a Medium Dose (Experimental): T-DM1 resistant/refractory (R/R) patients in the medium dose treatment group
  Interventions: Drug: DS-8201a
- DS-8201a High Dose (Experimental): T-DM1 resistant/refractory (R/R) patients in the high dose treatment group
  Interventions: Drug: DS-8201a
- Exploratory Arm (Other): In Part 2b- Continuation Stage, about 10 T-DM1 Intolerant patients will receive the DS-8201a recommended dose (RD) as an exploratory arm
  Interventions: Drug: DS-8201a

INTERVENTIONS:
Drug: DS-8201a — DS-8201a is sterile lyophilized powder reconstituted into a sterile aqueous solution (100 mg/5 mL) to be administered as low, medium and high intravenous (IV) doses for Part 1 of the trial. The dose for Part 2 will be determined based on results from Part 1.
  Other Names: Experimental product

SUMMARY:
Some human epidermal growth factor receptor 2 (HER-2) breast cancer patients do not respond or become resistant to current treatment. DS-8201a is a new experimental product that is a combination of an antibody and a drug. It has not yet been approved for use. DS-8201a may slow down tumor growth. This might improve outcomes for these patients.

ELIGIBILITY:
Inclusion Criteria:

* Men or women the age of majority in their country
* Has pathologically documented breast cancer that:

  1. is unresectable or metastatic
  2. has HER2 positive expression confirmed per protocol
* Has an adequate tumor sample
* Has at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Has protocol-defined adequate cardiac, renal and hepatic function
* Agrees to follow protocol-defined method(s) of contraception

Exclusion Criteria:

* Has a medical history of myocardial infarction, symptomatic congestive heart failure (CHF) (NYHA classes II-IV), unstable angina or serious cardiac arrhythmia
* Has a corrected QT interval (QTc) prolongation to > 450 millisecond (ms) in males and > 470 ms in females
* Has a medical history of clinically significant lung disease
* Is suspected to have certain other protocol-defined diseases based on imaging at screening period
* Has history of any disease, metastatic condition, drug/medication use or other condition that might, per protocol or in the opinion of the investigator, compromise:

  1. safety or well-being of the participant or offspring
  2. safety of study staff
  3. analysis of results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2017-08-25 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2024-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (99):
- United States (36):
  - Alaska Urological Institute dba Alaska Clinical Research Center, Anchorage, Alaska
  - Arizona Oncology Associates, Tucson, Arizona
  - The Regents of the University of California, Los Angeles, California
  - Sharp Clinical Oncology Research, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Sansum Clinic, Santa Barbara, California
  - Innovative Clinical Research Institute, LLC, Whittier, California
  - Sylvester Comprehensive Cancer Center - Deerfield Beach, Boca Raton, Florida
  - Specialist Global Research, Hialeah, Florida
  - Miami Cancer Institute at Baptist Health, Inc., Miami, Florida
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Straub Medical Center, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville Research Foundation, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - North Shore Hematology Oncology Associates PC DBA NY Cancer and Blood Specialists, East Setauket, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Aultman Hospital Cancer Center, Canton, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - St Francis Hospital, Greenville, South Carolina
  - Accurate Clinical Research, Baytown, Texas
  - Texas Oncology, P.A., Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The Methodist Hospital Research Institute, Houston, Texas
  - Texas Oncology, P.A. - Longview, Tyler, Texas
  - The University of Texas Health Science Center at Tyler, Tyler, Texas
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Providence Regional Medical Center - Everett, Everett, Washington
- Belgium (5):
  - Imeldaziekenhuis, Bonheiden
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Leuven, Leuven
  - CHU Sart Tilman, Liège
  - AZ Sint-Maarten, Mechelen
- University of Calgary, Calgary, Alberta, Canada
- France (15):
  - Institut Sainte Catherine, Avignon
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - Centre Georges François Leclerc, Dijon
  - CHU Bordeaux - Hôpital Saint André, Gironde
  - CH de la Rochelle - Hopital St Louis, La Rochelle
  - Clinique Victor Hugo - Centre Jean Bernard, Le Mans
  - Hôpital Nord - CHU Marseille, Marseille
  - Institut Régional du Cancer de Montpellier, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Hôpital Saint-Louis - Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CRLCC Eugene Marquis, Rennes
  - Hôpital d'Instruction des Armees Begin, Saint-Mandé
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Italy (6):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo), Monza
  - Ospedale degli Infermi, Rimini
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Torrette
- Japan (11):
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - Toranomon Hospital, Minatoku, Tokyo-To
  - Aichi Cancer Center Hospital, Aichi
  - National Cancer Center Hospital East, Chiba
  - NHO Kyushu Cancer Center, Fukuoka
  - Hakuaikai Sagara Hospital, Kagoshima
  - Kanagawa Cancer Center, Kanagawa
  - Kindai University Hospital, Osaka
  - National Cancer Center Hospital, Tokyo
  - St. Luke's International Hospital, Tokyo
  - Cancer Institute Hospital of JFCR, Tokyo
- South Korea (8):
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (11):
  - Hospital Infanta Cristina, Badajoz
  - Hospital Universitari Quiron Dexeus, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals, Barcelona
  - Hospital Quiron Barcelona, Barcelona
  - MD Anderson Cancer Centre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Virgen Macarena, Seville
  - Instituto Valenciano de Oncologia IVO, Valencia
- United Kingdom (6):
  - Derriford Hospital, Plymouth, Devon
  - Queen Mary University of London, London, Greater London
  - University College London Hospitals, London, Greater London
  - Western General Hospital, Edinburgh, Lothian Region
  - Nottingham University Hospitals City Campus, Nottingham, Nottinghamshire
  - Royal Surrey County Hospital, Guildford, Surrey

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Dunton K, Vondeling G, Hancock E, Petrou M, Burn O, Paine A. Methods for Estimating Long-Term Outcomes for Trastuzumab Deruxtecan in HER2-Positive Unresectable or Metastatic Breast Cancer After Two or More Anti-HER2 Therapies. Target Oncol. 2022 Nov;17(6):655-663. doi: 10.1007/s11523-022-00923-9. Epub 2022 Nov 7. PMID 36342619
- [Derived] Rugo HS, Bianchini G, Cortes J, Henning JW, Untch M. Optimizing treatment management of trastuzumab deruxtecan in clinical practice of breast cancer. ESMO Open. 2022 Aug;7(4):100553. doi: 10.1016/j.esmoop.2022.100553. Epub 2022 Aug 11. PMID 35964548
- [Derived] Bardia A, Harnden K, Mauro L, Pennisi A, Armitage M, Soliman H. Clinical Practices and Institutional Protocols on Prophylaxis, Monitoring, and Management of Selected Adverse Events Associated with Trastuzumab Deruxtecan. Oncologist. 2022 Aug 5;27(8):637-645. doi: 10.1093/oncolo/oyac107. PMID 35642907
- [Derived] Modi S. Trastuzumab deruxtecan in previously treated HER2-positive metastatic breast cancer: Plain language summary of the DESTINY-Breast01 study. Future Oncol. 2021 Sep 1;17(26):3415-3423. doi: 10.2217/fon-2021-0427. Epub 2021 Jul 15. PMID 34263665
- [Derived] Yin O, Iwata H, Lin CC, Tamura K, Watanabe J, Wada R, Kastrissios H, AbuTarif M, Garimella T, Lee C, Zhang L, Shahidi J, LaCreta F. Exposure-Response Relationships in Patients With HER2-Positive Metastatic Breast Cancer and Other Solid Tumors Treated With Trastuzumab Deruxtecan. Clin Pharmacol Ther. 2021 Oct;110(4):986-996. doi: 10.1002/cpt.2291. Epub 2021 Jun 10. PMID 33999422
- [Derived] Modi S, Saura C, Yamashita T, Park YH, Kim SB, Tamura K, Andre F, Iwata H, Ito Y, Tsurutani J, Sohn J, Denduluri N, Perrin C, Aogi K, Tokunaga E, Im SA, Lee KS, Hurvitz SA, Cortes J, Lee C, Chen S, Zhang L, Shahidi J, Yver A, Krop I; DESTINY-Breast01 Investigators. Trastuzumab Deruxtecan in Previously Treated HER2-Positive Breast Cancer. N Engl J Med. 2020 Feb 13;382(7):610-621. doi: 10.1056/NEJMoa1914510. Epub 2019 Dec 11. PMID 31825192

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met all of the inclusion and none of the exclusion criteria were enrolled and randomized to treatment (Part 1) or received DS-8201a at the recommended dose (Part 2).
Pre-assignment Details: In Part 1, participants were randomized 1:1:1 to either 5.4 mg/kg, 6.4 mg/kg, or 7.4 mg/kg dose of DS-8201a. Two doses randomized 1:1 (5.4 or 6.4 mg/kg) were further evaluated. In Part 2, all T-DM1 resistant refractory participants (cohort 2a) or T-DM1 intolerant (cohort 2b) received DS-8201a at the recommended dose.
Groups:
- Part 1: DS-8201a Low Dose: T-DM1 resistant/refractory (R/R) participants randomized to receive DS-8201a low dose (5.4 mg/kg) in the pharmacokinetic (PK) and dose-finding phases.
- Part 1: DS-8201a Medium Dose: T-DM1 resistant/refractory (R/R) participants randomized to receive DS-8201a medium dose (6.4 mg/kg) in the pharmacokinetic (PK) and dose-finding phases.
- Part 1: DS-8201a High Dose: T-DM1 resistant/refractory (R/R) participants randomized to receive DS-8201a high dose (7.4 mg/kg) in the pharmacokinetic (PK) and dose-finding phase.
- Part 2a: DS-8201a Low Dose: All T-DM1 resistant/refractory (R/R) participants who were treated at the recommended (5.4 mg/kg) dose in Part 2a in the continuation phase.
- Part 2b (Exploratory): DS-8201a Low Dose: All participants who were previously treated with T-DM1 and were randomized to receive DS8201a low dose (5.4 mg/kg) in Part 2b in the continuation phase.
Period: Overall Study
Arm/Group | Part 1: DS-8201a Low Dose | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 2a: DS-8201a Low Dose | Part 2b (Exploratory): DS-8201a Low Dose
Started | 50 | 48 | 21 | 130 | 4
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 50 | 48 | 21 | 130 | 4
Not completed — Progressive Disease | 24 | 23 | 11 | 66 | 1
Not completed — Adverse Event | 14 | 13 | 9 | 22 | 2
Not completed — Withdrawal by Subject | 5 | 4 | 0 | 8 | 1
Not completed — Physician Decision | 1 | 1 | 1 | 7 | 0
Not completed — Death | 1 | 1 | 0 | 6 | 0
Not completed — Study Terminated by Sponsor | 3 | 1 | 0 | 7 | 0
Not completed — Other | 2 | 5 | 0 | 14 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part 1: DS-8201a High Dose: T-DM1 resistant/refractory (R/R) participants randomized to receive DS-8201a high dose (7.4 mg/kg) in the pharmacokinetic (PK) and dose-finding phases.
- Total: Total of all reporting groups
Arm/Group | Part 1: DS-8201a Low Dose | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 2a: DS-8201a Low Dose | Part 2b (Exploratory): DS-8201a Low Dose | Total
Number analyzed (Participants) | 50 | 48 | 21 | 130 | 4 | 253
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 35 | 33 | 16 | 101 | 4 | 189
  >=65 years | 15 | 15 | 5 | 29 | 0 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.9 (11.3) | 55.8 (13.0) | 54.4 (10.5) | 55.4 (11.9) | 49.8 (9.2) | 55.8 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 48 | 21 | 130 | 4 | 253
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1 | 2
  Asian | 22 | 22 | 12 | 47 | 1 | 104
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 2 | 0 | 1 | 1 | 1 | 5
  White | 24 | 23 | 8 | 76 | 1 | 132
  More than one race | 1 | 1 | 0 | 2 | 0 | 4
  Unknown or Not Reported | 0 | 1 | 0 | 4 | 0 | 5
Region of Enrollment [Number; unit: participants]
  South Korea | 7 | 7 | 0 | 25 | 1 | 40
  Belgium | 0 | 2 | 0 | 7 | 0 | 9
  United States | 15 | 14 | 10 | 36 | 2 | 77
  Japan | 16 | 15 | 11 | 14 | 0 | 56
  Italy | 0 | 1 | 0 | 8 | 1 | 10
  United Kingdom | 0 | 0 | 0 | 12 | 0 | 12
  France | 2 | 1 | 0 | 17 | 0 | 20
  Spain | 10 | 8 | 0 | 11 | 0 | 29

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate as Confirmed by Independent Central Review Following Intravenous Administration of 5.4 mg/kg DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: The number of participants with objective response was assessed every six weeks from Cycle 1 Day 1 through discontinuation of treatment, by independent central imaging facility review based on RECIST version 1.1.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Objective response rate (ORR) was assessed in the Enrolled Analysis Set.at data cut-off date of 21 March 2019
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 and Part 2a: DS-8201a Low Dose: All T-DM1 resistant/refractory (R/R) participants who were treated in Part 1 or Part 2a at the recommended (5.4 mg/kg) dose.
- Part 1 + Part 2a + Part 2b: DS-8201a Low Dose: All participants who were previously treated with T-DM1 and were randomized to receive DS8201a low dose (5.4 mg/kg) in Part 1 or Part 2a or Part 2b.
Arm/Group | Part 1 and Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 180 | 184
Participants | 109 | 111

2. Secondary Outcome: Objective Response Rate as Confirmed By the Investigator Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: The number of participants with objective response is assessed every six weeks from Cycle 1 Day 1 through discontinuation of treatment. Investigator-assessed objective response rate (ORR) was defined as the proportion of participants who achieved a best overall response of complete response or partial response based on local radiologists/investigators' tumor assessments.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Objective response rate (ORR) was assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 and Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose
Number analyzed (Participants) | 180 | 184 | 48 | 21
Participants | 116 | 118 | 37 | 18

3. Secondary Outcome: Best Overall Tumor Response as Confirmed By the Investigator Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: Best overall tumor response was defined as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) by the investigator based on RECIST v1.1. Participants who were non-evaluable (NE) are also reported.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Best overall tumor response was assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Count of Participants; unit: Participants
Groups:
- Part 1 + Part 2a: DS-8201a Low Dose: All T-DM1 resistant/refractory (R/R) participants who were treated at the recommended (5.4 mg/kg) dose in Part 1 or Part 2a.
Arm/Group | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 1 + Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 48 | 21 | 180 | 184
Participants
  Complete response | 3 | 0 | 4 | 6
  Partial response | 34 | 18 | 112 | 112
  Stable disease | 10 | 3 | 59 | 61
  Progressive disease | 0 | 0 | 4 | 4
  Non-evaluable | 1 | 0 | 1 | 1

4. Secondary Outcome: Disease Control Rate and Clinical Benefit Rate as Confirmed by Independent Central Review Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: Number of participants with controlled disease and who received clinical benefit from treatment as assessed by independent central review. DCR was defined as the proportion of participants who achieved a best overall response of complete response, partial response, or stable disease. CBR was defined as the proportion of participants who achieved a best overall response of complete response or partial response or more than 6 months of stable disease.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Disease control rate (DCR) and clinical benefit rate (CBR) were assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 1 + Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 48 | 21 | 180 | 184
Participants
  Disease control rate | 47 | 21 | 175 | 179
  Clinical benefit rate | 41 | 20 | 127 | 130

5. Secondary Outcome: Duration of Response (Complete Response or Partial Response) as Confirmed by Independent Central Review Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: The estimated duration of confirmed response (complete response [CR] or partial response [PR]) was assessed by independent central review. Duration of response was defined as the time interval between the date of first documentation of objective response (CR or PR) and the date of the first objective documentation of disease progression or death due to any cause.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Participants with CR or PR were analyzed. Estimated duration of response was assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 1 + Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 33 | 17 | 109 | 111
months | NA [8.3 to NA] — There were not enough events to estimate a standard error for the median survival time. | 6.0 [4.8 to 8.3] | NA [NA to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. | NA [NA to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event.

6. Secondary Outcome: Progression-Free Survival Estimate As Confirmed by Independent Central Review Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: The point estimate of progression-free survival (PFS) is reported. PFS was defined as the time interval between the date of randomization/registration and the first documentation of disease progression or death due to any cause.
Time Frame: at least 6 months after last participant enrolled received first dose up to 19 months (data cut off)
Population: Progression-free survival was assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 1 + Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 48 | 21 | 180 | 184
months | NA [NA to NA] — Lack of a median value is due to less than 50% of the participants experiencing the event. | 9.5 [7.4 to 13.2] | NA [10.6 to NA] — There were not enough events to estimate a standard error for the median survival time. | NA [10.6 to NA] — There were not enough events to estimate a standard error for the median survival time.

7. Secondary Outcome: Percent Change From Baseline in Sum of Diameters Over Time as Determined by Independent Central Review Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Enrolled Analysis Set)
Description: Best percent change in sum of diameters of measurable tumors was based on RECIST 1.1. The best percent change was defined as the percent change in the smallest sum of diameters from all post-baseline tumor assessments, taking as reference the baseline sum of diameters.
Time Frame: Baseline up to Week 6, 12, 18, 24, 30, 36 post dose
Population: Best percent change from baseline in sum of diameters was assessed in the Enrolled Analysis Set at data cut-off date of 21 March 2019.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 1 + Part 2a: DS-8201a Low Dose | Part 1 + Part 2a + Part 2b: DS-8201a Low Dose
Number analyzed (Participants) | 48 | 21 | 180 | 184
Percent change from baseline
  Baseline to Week 6: number analyzed (Participants) | 43 | 21 | 164 | 167
  Baseline to Week 6 | -26.2 (18.3) | -32.9 (25.4) | -26.9 (21.6) | -26.9 (22.5)
  Baseline to Week 12: number analyzed (Participants) | 40 | 21 | 152 | 154
  Baseline to Week 12 | -39.6 (22.7) | -43.6 (28.1) | -39.9 (24.5) | -40.1 (24.9)
  Baseline to Week 18: number analyzed (Participants) | 37 | 19 | 136 | 138
  Baseline to Week 18 | -50.1 (22.1) | -58.5 (29.4) | -44.4 (27.8) | -44.9 (28.0)
  Baseline to Week 24: number analyzed (Participants) | 31 | 17 | 124 | 125
  Baseline to Week 24 | -56.3 (22.1) | -61.9 (32.0) | -49.2 (30.6) | -49.3 (30.5)
  Baseline to Week 30: number analyzed (Participants) | 30 | 15 | 80 | 81
  Baseline to Week 30 | -59.1 (26.1) | -63.9 (32.2) | -51.2 (29.2) | -51.5 (29.2)
  Baseline to Week 36: number analyzed (Participants) | 24 | 9 | 46 | 46
  Baseline to Week 36 | -61.0 (26.7) | -54.6 (32.2) | -55.5 (29.9) | -55.5 (29.9)
  Best percent change from baseline: number analyzed (Participants) | 43 | 21 | 166 | 169
  Best percent change from baseline | -59.5 (28.2) | -65.3 (27.7) | -50.5 (28.3) | -50.6 (28.8)

8. Secondary Outcome: Overall Summary of Treatment-emergent Adverse Events (TEAEs) Following Intravenous Administration of DS-8201a in Participants With Metastatic Breast Cancer (Safety Analysis Set)
Description: TEAEs were assessed by severity and seriousness according to unique criteria. Severity described the intensity of an event and was graded using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03, where Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL); Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL; Grade 4: Life-threatening consequences; urgent intervention indicated; and Grade 5: Death related to AE. Serious TEAEs were defined as any untoward medical occurrence that at any dose results in death, is life threatening, requires inpatient hospitalization, or causes prolongation of existing hospitalization.
Time Frame: Day 0 to Day 47 post last dose
Population: Adverse event data were assessed in the Safety Analysis Set t data cut-off date of 21 March 2019.
Measure: Count of Participants; unit: Participants
Groups:
- Part 2a: DS-8201a Low Dose: All T-DM1 resistant/refractory (R/R) participants who were treated at the recommended (5.4 mg/kg) dose in the continuation phase.
- Part 2b (Exploratory): DS-8201a Low Dose: All participants who were T-DM1 intolerant and treated at the recommend dose (5.4 mg/kg) in the continuation phase.
Arm/Group | Part 1: DS-8201a Low Dose | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 2a: DS-8201a Low Dose | Part 2b (Exploratory): DS-8201a Low Dose
Number analyzed (Participants) | 50 | 48 | 21 | 130 | 4
Participants
  Any TEAE | 50 | 48 | 21 | 129 | 4
  Drug-related TEAEs | 50 | 47 | 21 | 128 | 4
  Drug-related TEAEs of CTCAE ≥Grade 3 | 26 | 32 | 16 | 48 | 3
  Any serious TEAE | 11 | 6 | 8 | 25 | 0
  Drug-related serious TEAEs | 6 | 4 | 5 | 10 | 0
  TEAEs associated with drug discontinuation | 6 | 6 | 8 | 8 | 1
  Related TEAEs associated with drug discontinuation | 6 | 6 | 8 | 7 | 1
  TEAEs associated with dose reduction | 13 | 19 | 11 | 21 | 3
  Drug-related TEAEs associated with dose reduction | 11 | 18 | 11 | 20 | 3
  TEAEs associated with dose interruption | 19 | 16 | 12 | 36 | 2
  Related TEAEs associated with drug interruption | 17 | 13 | 11 | 29 | 2
  TEAEs associated with death | 1 | 1 | 2 | 8 | 0
  Drug-related TEAEs associated with death | 0 | 0 | 1 | 2 | 0

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected from Day 0 through Day 47 post last dose of study drug.
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event (AE) that occurred, having been absent before the first dose of study drug, or had worsened in severity or seriousness after the initiating the study drug until 47 days after last dose of the study drug.
Groups:
- Part 2b (Exploratory): DS-8201a Low Dose: All participants who were T-DM1 intolerant and treated at the recommend dose (5.4 mg/kg) in Part 2b in the continuation phase.
Arm/Group | Part 1: DS-8201a Low Dose | Part 1: DS-8201a Medium Dose | Part 1: DS-8201a High Dose | Part 2a: DS-8201a Low Dose | Part 2b (Exploratory): DS-8201a Low Dose
All-Cause Mortality (participants affected / at risk) | 33/50 | 30/48 | 18/21 | 86/130 | 3/4
Serious Adverse Events (participants affected / at risk) | 14/50 | 11/48 | 8/21 | 42/130 | 1/4
Other Adverse Events (participants affected / at risk) | 50/50 | 48/48 | 21/21 | 129/130 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part 1: DS-8201a Low Dose (N=50) | Part 1: DS-8201a Medium Dose (N=48) | Part 1: DS-8201a High Dose (N=21) | Part 2a: DS-8201a Low Dose (N=130) | Part 2b (Exploratory): DS-8201a Low Dose (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Hematuria (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Shock haemorrhagic (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 | 3 (3) | 0 (0) | 3 (4) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Abdominal abscess (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 | 0
Disease progression (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Pain (General disorders) | 0 | 0 | 1 (1) | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pyelonephritis (Infections and infestations) | 1 (1) | 0 | 0 | 1 (4) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 3 (3) | 0 | 0 | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 (1) | 0 (0) | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 1 (1) | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0)
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Pneumonitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0)
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1 (1) | 0 (0) | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0 | 0
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 (3) | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 (3) | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 (2) | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0
Epilepsy (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 (1) | 0 | 0 | 0 | 0
Genital hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (20) | 0 | 1 (1) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 1 (1) | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 (2) | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Gastric varices (Gastrointestinal disorders) | 1 (2) | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 (1) | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 (1) | 0 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0/0 (0) | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary valve disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dehiscence (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: DS-8201a Low Dose (N=50) | Part 1: DS-8201a Medium Dose (N=48) | Part 1: DS-8201a High Dose (N=21) | Part 2a: DS-8201a Low Dose (N=130) | Part 2b (Exploratory): DS-8201a Low Dose (N=4)
Neutropenia (Blood and lymphatic system disorders) | 9 (37) | 7 | 5 | 13 | 1
Lymphopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 10 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 11 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 7 | 1
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 5 | 1
Dry eye (Eye disorders) | 4 | 7 | 7 | 18 | 0
Keratitis (Eye disorders) | 2 | 3 | 3 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 3 | 4 | 0 | 0
Visual impairment (Eye disorders) | 1 | 2 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 38 | 40 | 13 | 102 | 3
Vomiting (Gastrointestinal disorders) | 23 | 21 | 8 | 61 | 2
Constipation (Gastrointestinal disorders) | 16 | 19 | 10 | 50 | 1
Diarrhea (Gastrointestinal disorders) | 16 | 16 | 5 | 41 | 1
Stomatitis (Gastrointestinal disorders) | 12 | 16 | 4 | 17 | 2
Dyspepsia (Gastrointestinal disorders) | 4 | 5 | 0 | 28 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 4 | 3 | 20 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 4 | 2 | 11 | 1
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 0 | 13 | 0
Hemorrhoids (Gastrointestinal disorders) | 5 | 2 | 1 | 7 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 2 | 4 | 0
Ascites (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 3 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0
Fatigue (General disorders) | 22 | 25 | 11 | 70 | 2
Asthenia (General disorders) | 9 | 9 | 0 | 16 | 1
Pyrexia (General disorders) | 5 | 14 | 5 | 16 | 0
Mucosal inflammation (General disorders) | 1 | 4 | 0 | 16 | 0
Odema peripheral (General disorders) | 4 | 8 | 0 | 13 | 2
Malaise (General disorders) | 3 | 4 | 5 | 2 | 0
Urinary tract infection (Infections and infestations) | 6 | 4 | 3 | 16 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5 | 1 | 18 | 0
Nasopharyngitis (Infections and infestations) | 7 | 3 | 3 | 13 | 0
Cystitis (Infections and infestations) | 3 | 2 | 1 | 3 | 1
Cellulitis (Infections and infestations) | 3 | 1 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 0 | 0 | 1 | 1
Influenza (Infections and infestations) | 0 | 3 | 1 | 3 | 0
Conjunctivitis (Infections and infestations) | 0 | 4 | 1 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 3 | 0 | 0 | 0
Infusion-related reaction (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 16 | 19 | 13 | 25 | 0
White blood cell count decreased (Investigations) | 14 | 17 | 13 | 22 | 0
Platelet count decreased (Investigations) | 11 | 14 | 7 | 20 | 1
Aspartate aminotransferase increased (Investigations) | 9 | 7 | 5 | 19 | 0
Alanine aminotransferase increased (Investigations) | 8 | 7 | 5 | 14 | 0
Lymphocyte count decreased (Investigations) | 4 | 7 | 2 | 16 | 0
Weight decreased (Investigations) | 6 | 7 | 5 | 9 | 1
Blood bilirubin increased (Investigations) | 4 | 3 | 5 | 11 | 0
Blood alkaline phosphatase increased (Investigations) | 3 | 6 | 6 | 9 | 0
Electrocardiogram QT prolonged (Investigations) | 6 | 0 | 1 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 4 | 0 | 3 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 6 | 1 | 7 | 0
Troponin I increased (Investigations) | 3 | 0 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 1 | 0 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 17 | 22 | 6 | 43 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 3 | 4 | 15 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3 | 4 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 3 | 18 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 8 | 1 | 16 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0 | 13 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1 | 12 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 9 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0
Headache (Nervous system disorders) | 8 | 13 | 2 | 32 | 2
Dysgeusia (Nervous system disorders) | 5 | 7 | 1 | 8 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 5 | 2 | 13 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 1 | 2 | 8 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 5 | 5 | 7 | 0
Anxiety (Psychiatric disorders) | 3 | 5 | 2 | 9 | 0
Dizziness (Psychiatric disorders) | 7 | 6 | 1 | 13 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 1 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 5 | 34 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 2 | 24 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 8 | 5 | 1 | 20 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 3 | 7 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 4 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 25 | 29 | 8 | 62 | 2
Rash (Skin and subcutaneous tissue disorders) | 5 | 8 | 1 | 16 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 1 | 9 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 8 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 4 | 0 | 10 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 20 (51) | 21 (68) | 10 (30) | 39 (139) | 1 (1)
Chills (General disorders) | 3 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 3 | 0 | 0 | 10 | 0
COVID-19 (Infections and infestations) | 3 | 4 | 0 | 8 | 0
Pneumonia (Infections and infestations) | 3 | 3 | 1 | 0 | 0
Troponin increased (Investigations) | 3 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 5 | 4 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 5 | 4 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0 | 3 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 3 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 3 | 0 | 0 | 2 | 1
Lymphoedema (Vascular disorders) | 3 | 0 | 0 | 7 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 3 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 4 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 1
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 9 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 7 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03248492/Prot_SAP_000.pdf